CLINICAL TRIAL: NCT01417065
Title: Phase 0 Trial Evaluating the Effect of Temsirolimus on Known Pharmacodynamic Targets
Brief Title: Temsirolimus In Phase 0
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0259; NCI-2011-02799 (Registry Identifier: NCI CTRP); 2K12CA088084-12 (NIH)
Record Dates: First submitted 2011-08-12; First posted 2011-08-16 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Advanced Cancer
Keywords: Cancer; mTOR inhibitor Temsirolimus; Torisel; CCI-779; pharmacodynamic targets
MeSH Terms: conditions — Neoplasms | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temsirolimus (Experimental): Starting dose 0.02 mg intravenous administered once.
  Interventions: Drug: Temsirolimus

INTERVENTIONS:
Drug: Temsirolimus — Starting dose will be 0.02 mg intravenous administered once on Day 1 over 60 minutes.
  Other Names: CCI-779; Torisel

SUMMARY:
The goal of this clinical research trial is to study the effects of the FDA-approved drug, temsirolimus, using a new type of clinical study design called a "Phase 0." This type of study may be able to predict if a drug can affect cancer and may be able to prevent potentially useful study drugs from being discarded before they are fully tested.

The purpose of the study is not to treat the cancer, but to help improve general cancer treatment knowledge.

DETAILED DESCRIPTION:
Study Drug:

Temsirolimus is designed to block the growth of cancer cells, which may cause the cancer cells to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive temsirolimus by vein over about 60 minutes on Day 1.

You will be assigned to a dose level of temsirolimus based on when you join this study. Up to 5 dose levels of temsirolimus will be tested. Up to 3 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, until the drug is found to affect the enzyme that was tested for at screening.

Study Visits:

At each study visit, you will be asked about any drugs you may be taking and about any side effects you may be having.

On Day 1:

-Blood (about 2 teaspoons each time) will be drawn before you receive the study drug and 5 times over the 24 hours after you receive the study drug for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points.

Blood (about 4 teaspoons each time) will be drawn for pharmacodynamic (PD) testing. PD testing measures how the level of study drug in your body may affect the disease. This blood will be drawn at 1 or more of the following times, but if the doctor thinks it is needed, blood will be drawn at 2 or all 3 of the following times:

* At 4 hours (+/- 2 hours) after the dose
* At 24 hours (+/- 3 hours) after the dose
* At 72 hours (+/- 24 hours) after the dose

After the blood for PD testing has been tested and the tests show that the study drug may be causing changes to the tumor cells in at least 2 out of 3 participants, future participants will have tumor tissue collected before and after dosing for testing. Leftover tissue from an earlier biopsy can be used instead of a fresh biopsy before dosing, if it is available.

Length of Study:

You will be on study for up to 4 days. You will be taken off study early if you have intolerable side effects.

Because it takes 4 days for temsirolimus to be completely processed by the body, you will not be able to begin receiving drugs in any other study until 4 days after the dose.

This is an investigational study. Temsirolimus is FDA approved and commercially available for the treatment of advanced renal cancer. Its use in other types of cancer is investigational.

Up to 30 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic cancer, preferably with tumor easily accessible for biopsy.
2. Patients should be at least four weeks or 5 half lives from the last day of chemotherapy, antibody or other biological therapy, whichever is shorter.
3. Patients should preferably be undergoing screening for 2007-0668, 2008-0384, 2008-0425, and 2008-0827 (currently active Phase I trials involving temsirolimus). However, patients may also be allowed on protocol if they are undergoing screening for any study.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with a known hypersensitivity to any of the components or metabolites of the drug products.
3. Patients with a known bleeding diathesis which would prevent safely obtaining a biopsy if a biopsy is indicated.
4. Patients who are less than 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-08; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Participants' Pharmacodynamic (PD) Responses | Blood drawn at 4 hours (+/- 2 hours) after study drug
  PD response, significant S6 Kinase 1 (S6K1) inhibition, is defined at both the patient level and the dose level, 1) as compared with baseline, at least 50% reductions of S6K1 after treatment (biological criterion); 2) differences in log transformed S6K1 activity between post-treatment and baseline should be greater than threshold of 1.8 times standard deviation (SD) of baseline, which yields a 90% statistical confidence that it is not due to chance variation (statistical criterion).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Karp, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org